CLINICAL TRIAL: NCT06661785
Title: Interlocking Polyetheretherketone Patient-Specific Implants for Orbital Floor Reconstruction
Brief Title: Interlocking Polyetheretherketone Implants for Orbital Floor Reconstruction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Maram Nashaat Breshah, Lecturer of Oral & Maxillofacial Surgery, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #R-OS-12-22-3
Record Dates: First submitted 2024-10-22; First posted 2024-10-28 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2024-10

CONDITIONS: Large Orbital Floor Fracture
Keywords: orbital reconstruction; Interlocking PEEK; Patient specific implant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interlocking polyetheretherketone patient specific implant for orbital floor reconstruction (Experimental): This study is conducted on twenty two patients with unilateral large orbital floor fracture reconstructed with interlocking polyetheretherketone patient specific implant
  Interventions: Procedure: large orbital floor fracture

INTERVENTIONS:
Procedure: large orbital floor fracture — Twenty two patients with large orbital floor fracture will be reconstructed with interlocking polyetheretherketone patient-specific implant

SUMMARY:
Patients with large orbital floor fracture were reconstructed with interlocking polyetheretherketone patient-specific implant and will be evaluated clinically and radiographically

DETAILED DESCRIPTION:
Twenty two patients with large orbital floor fracture will be included in this study. Patients will be received, examined and managed at the Oral & Maxillofacial Surgery Department, Faculty of Dentistry, Tanta University. Full clinical examination and radiographic examination using multi axial C.T Scan for proper diagnosis and treatment planning. DICOM files will be imported into surgical planning software and used for fabrication of interlocking polyetheretherketone patient specific implant which will be ready for sterilization and insertion. After written informed consent from the patient, the surgery will be done under G.A, either infraorbital or transconjunctival incision will be done according to the case. Follow up: All patients will be examined clinically for hypoglobus, enophthalmos, ocular motility and diplopia during 2nd week, 1st month and 6 months & radiographically for orbital volume immediately and 6 months postoperatively

ELIGIBILITY:
Inclusion Criteria:

* Patients with large orbital blow out fracture either isolated or combined with other fracture
* Patients willing for surgical operation and follow up
* Patients with no contraindications for surgical intervention

Exclusion Criteria:

* Patients who are not fit for G.A
* Uncooperative patients

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2025-11-02 (Estimated)

PRIMARY OUTCOMES:
Hypoglobus | 2 weeks
  It is the downward displacement of the eyeball of affected eye. It is measured by drawing imaginary line horizontally across the patient's inter-pupillary axis and determine if the pupil of the affected eye is lower or not
Enophthalmos | 2 weeks
  It is defined as the posterior displacement of the eyeball within the orbit. It was measured by the aid of exophthalmometer. Assessment is consisting of four grades as follow:
  grade 0:no enophthalmos grade 1:mild enophthalmos(less than 1 mm) grade 2:moderate enophthalmos(from 1 to 2 mm) grade 3:severe enophthalmos(over 2 mm)
Orbital volume | 2 weeks
  C.T. images of the patient are imported in DICOM format into the automatic orbital analysis software and the orbital volume of both orbital cavities are measured
Ocular motility | 2 weeks
  It is done by asking the patient to follow a moving target into the diagnostic positions of gaze, observing the extent of movement of each eye. The amount of limitation of movement is classified as:
  grade 1:slight limitation grade 2:moderate limitation grade 3:marked limitation grade 4:no movement
Diplopia | 2 weeks
  It is defined as perception of two images of the same object in visual space. It is assessed if it is present in primary position of gaze or in secondary position of gaze

SECONDARY OUTCOMES:
Hypoglobus | 6 months
  It is the downward displacement of the eyeball of affected eye. It is measured by drawing imaginary line horizontally across the patient's inter-pupillary axis and determine if the pupil of the affected eye is lower or not
Enophthalmos | 6 months
  It is defined as the posterior displacement of the eyeball within the orbit. It was measured by the aid of exophthalmometer. Assessment is consisting of four grades as follow: grade 0:no enophthalmos grade 1:mild enophthalmos(less than 1 mm) grade 2:moderate enophthalmos(from 1 to 2 mm) grade 3:severe enophthalmos(over 2 mm)
Orbital volume | 6 months
  C.T. images of the patient are imported in DICOM format into the automatic orbital analysis software and the orbital volume of both orbital cavities are measured
Ocular motility | 6 months
  It is done by asking the patient to follow a moving target into the diagnostic positions of gaze, observing the extent of movement of each eye. The amount of limitation of movement is classified as: grade 1:slight limitation grade 2:moderate limitation grade 3:marked limitation grade 4:no movement
Diplopia | 6 months
  It is defined as perception of two images of the same object in visual space. It is assessed if it is present in primary position of gaze or in secondary position of gaze

CONTACTS AND LOCATIONS:
Overall Officials: Maram N Breshah, Lecturer, Principal Investigator — Tanta University, Egypt; Rafic R Beder, Prof, Principal Investigator — Tanta University, Egypt
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No